CLINICAL TRIAL: NCT00516217
Title: A Phase II Study of Galiximab (Anti-CD80) for Patients With Relapsed/Refractory Hodgkin Lymphoma
Brief Title: Galiximab in Treating Patients With Relapsed or Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-50602; U10CA031946 (NIH); CALGB-50602; CDR0000561185 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Results first posted 2015-02-04 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; adult lymphocyte predominant Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — galiximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Galaximab (Experimental): Induction: 500 mg/m^2 by IV over 60 minutes days 1, 8, 15 & 22 Extended Induction: 500 mg/m^2 by IV every 4 weeks until disease progression or unacceptable toxicity
  Interventions: Biological: galiximab

INTERVENTIONS:
Biological: galiximab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as galiximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them.

PURPOSE: This phase II trial is studying how well galiximab works in treating patients with relapsed or refractory Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the response rate (complete and overall response) in patients with relapsed or refractory Hodgkin lymphoma (HL) treated with galiximab.

Secondary

* To assess the duration of response, progression-free survival, and overall survival of patients with relapsed or refractory HL.
* To assess the safety and tolerability of galiximab in patients with relapsed or refractory HL.
* To determine if FDG-PET correlates with outcome in patients with relapsed or refractory HL treated with galiximab.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive galiximab IV over 60 minutes on days 1, 8, 15, and 22 in month 1.
* Extended induction therapy: Patients receive galiximab IV over 60 minutes once every four weeks in the absence of disease progression or unacceptable toxicity.

Patients also undergo FDG-PET/CT imaging at baseline and at time of first restaging (within 7 days prior to week 8 treatment).

After completion of study treatment, patients are followed periodically for 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed classical Hodgkin lymphoma (HL):

  * Bone marrow biopsies as the sole means of diagnosis are not acceptable, but they may be submitted in conjunction with nodal biopsies
  * Fine needle aspirates are not acceptable
* Recurrent or refractory disease after at least two prior standard chemotherapy regimens
* Nodular lymphocyte predominant HL allowed
* Measurable disease must be present on either physical examination or imaging studies

  * Measurable disease is defined as any lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm
  * Evaluable or non-measurable disease alone is not acceptable including any of the following:

    * Bone lesions (lesions, if present, should be noted)
    * Bone marrow involvement (if present, this should be noted)
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
* Ineligible for a stem cell transplantation
* Patients eligible for CALGB-50502 should not be considered for this study
* No known CNS involvement

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 500/μL
* Platelet count ≥ 50,000/μL
* Creatinine ≤ 2.0 mg/dL
* Total bilirubin ≤ 2.0 mg/dL (no history of Gilbert Disease)
* AST ≤ 2.5 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study
* No known HIV infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered to ≤ grade 1 from all toxicities related to prior treatments
* At least 4 weeks since prior chemotherapy, radiotherapy, or biologic anticancer therapy
* Prior autologous and/or allogeneic stem cell transplantation allowed
* No prior anti-CD80 antibody
* No concurrent steroids, hormones, or other chemotherapeutic agents except for steroids given for adrenal failure and hormones administered for non-disease-related conditions (e.g., insulin for diabetes)

  * The use of dexamethasone and other steroidal antiemetics is prohibited unless to treat acute grade 3 or 4 monoclonal antibody-associated infusion reactions not responsive to transient discontinuation of antibody infusion or acetaminophen and diphenhydramine
  * Dexamethasone is also allowed for re-treatment after an infusion reaction

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2011-09 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Smith, MD, Study Chair — University of Chicago
Locations (56):
- United States (56):
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Danville Regional Medical Center, Danville, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2008 and January 2009, 30 patients were recruited.
Pre-assignment Details: One patient never received treatment and is excluded from all analyses.
Period: Overall Study
Arm/Group | Galaximab
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Galaximab
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 36 [22 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Overall response is defined as achievement of a complete response (CR) or partial response (PR) as defined by the Revised Response Criteria for Malignant Lymphoma.
  CR: complete disappearance of all detectable disease PR: >=50% decrease in the sum of the product of diameters of indicator lesions.
Time Frame: Duration of treatment (up to 10 years)
Measure: Number; unit: participants
Arm/Group | Galaximab
Number analyzed (Participants) | 29
participants | 3

2. Secondary Outcome: 12 Month Overall Survival Rate
Description: Percentage of patients who were alive at 12 months. The 12-month survival rate was estimated using the Kaplan Meier method.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Galaximab
Number analyzed (Participants) | 29
percentage of participants | 79 [59 to 90]

3. Secondary Outcome: 6 Month Progression Free Survival Rate
Description: Percentage of patients who were progression free at 6 months. The 6-month progression free rate was estimated using the Kaplan Meier method.
  Relapse was assessed by investigator according to Revised Response Criteria for Malignant Lymphoma. Progression required a appearance of any new lesion > 1.5 cm, at least 50% increase from nadir in the sum of products of involved nodes, or a 50% increase in the longest diameter of any single node.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Galaximab
Number analyzed (Participants) | 29
percentage of participants | 21 [8 to 37]

ADVERSE EVENTS:
Groups:
- Galaximab: Extended Induction: 500 mg/m^2 by IV every 4 weeks until disease progression or unacceptable toxicity
Arm/Group | Galaximab
Serious Adverse Events (participants affected / at risk) | 8/29
Other Adverse Events (participants affected / at risk) | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galaximab (N=29)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 (9)
Cardiac disorder (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (4)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (12)
Vomiting (Gastrointestinal disorders) | 4 (5)
Chills (General disorders) | 3 (5)
Edema limbs (General disorders) | 2 (3)
Facial pain (General disorders) | 1 (2)
Fatigue (General disorders) | 6 (14)
Fever (General disorders) | 6 (13)
General symptom (General disorders) | 1 (1)
Pain (General disorders) | 3 (4)
Autoimmune disorder (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Anal infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 3 (4)
Joint infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (7)
Alkaline phosphatase increased (Investigations) | 5 (10)
Aspartate aminotransferase increased (Investigations) | 4 (10)
Blood bilirubin increased (Investigations) | 2 (3)
Cardiac troponin T increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 2 (5)
Gamma-glutamyltransferase increased (Investigations) | 3 (7)
INR increased (Investigations) | 2 (4)
Leukocyte count decreased (Investigations) | 2 (3)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (4)
Neutrophil count decreased (Investigations) | 3 (5)
Platelet count decreased (Investigations) | 6 (14)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (6)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (10)
Serum albumin decreased (Metabolism and nutrition disorders) | 4 (11)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (9)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 4 (5)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (6)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 5 (7)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5)
Headache (Nervous system disorders) | 2 (4)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (5)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (3)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 3 (5)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galaximab (N=29)
Blood disorder (Blood and lymphatic system disorders) | 1 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 17 (33)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Cardiac pain (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (17)
Adrenal insufficiency (Endocrine disorders) | 1 (2)
Cushingoid (Endocrine disorders) | 1 (3)
Hypothyroidism (Endocrine disorders) | 2 (2)
Dry eye syndrome (Eye disorders) | 1 (10)
Flashing vision (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 6 (8)
Dry mouth (Gastrointestinal disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (14)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Gastric mucositis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (24)
Vomiting (Gastrointestinal disorders) | 5 (6)
Chills (General disorders) | 6 (8)
Edema limbs (General disorders) | 4 (15)
Fatigue (General disorders) | 24 (52)
Fever (General disorders) | 10 (13)
Localized edema (General disorders) | 2 (2)
Pain (General disorders) | 1 (2)
Anorectal infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (2)
Infection (Infections and infestations) | 1 (1)
Infectious colitis (Infections and infestations) | 1 (1)
Joint infection (Infections and infestations) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3)
Upper respiratory infection (Infections and infestations) | 2 (4)
Urinary tract infection (Infections and infestations) | 1 (3)
Bruising (Injury, poisoning and procedural complications) | 2 (5)
Alanine aminotransferase increased (Investigations) | 8 (13)
Alkaline phosphatase increased (Investigations) | 10 (20)
Aspartate aminotransferase increased (Investigations) | 6 (12)
Blood bilirubin increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 4 (5)
Gamma-glutamyltransferase increased (Investigations) | 1 (3)
Laboratory test abnormal (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 4 (7)
Lymphocyte count decreased (Investigations) | 9 (16)
Neutrophil count decreased (Investigations) | 2 (5)
Platelet count decreased (Investigations) | 15 (38)
Serum cholesterol increased (Investigations) | 2 (6)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (9)
Blood glucose increased (Metabolism and nutrition disorders) | 14 (27)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 7 (11)
Serum calcium decreased (Metabolism and nutrition disorders) | 6 (8)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (3)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 6 (11)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 6 (12)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (13)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Acoustic nerve disorder NOS (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 4 (6)
Neuralgia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (7)
Speech disorder (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (4)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Hemoglobin urine positive (Renal and urinary disorders) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (22)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (30)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (17)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (4)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (3)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.